CLINICAL TRIAL: NCT00263822
Title: A Randomized, Multicenter, Phase III Study of Erlotinib Versus Observation in Patients With no Evidence of Disease Progression After First Line, Platinum-Based Chemotherapy For High-Risk Ovarian Epithelial, Primary Peritoneal, or Fallopian Tube Cancer
Brief Title: Erlotinib or Observation in Treating Patients Who Have Undergone First-Line Chemotherapy for Ovarian Cancer, Peritoneal Cancer, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-55041; EORTC-55041; EUDRACT-2004-004333-34
Record Dates: First submitted 2005-12-07; First posted 2005-12-09 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; primary peritoneal cavity cancer; fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: erlotinib hydrochloride

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Sometimes after treatment, the tumor may not need additional treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether erlotinib is more effective than observation after first-line chemotherapy in treating patients with ovarian cancer, peritoneal cancer, or fallopian tube cancer.

PURPOSE: This randomized phase III trial is studying erlotinib to see how well it works compared to observation in treating patients who have undergone first-line chemotherapy for ovarian cancer, peritoneal cancer, or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the benefits, in terms of progression-free survival, of maintenance therapy comprising erlotinib vs observation in patients with responding or stable disease after first-line, platinum-based chemotherapy for high-risk stage I or stage II-IV ovarian epithelial, primary peritoneal, or fallopian tube cancer.

Secondary

* Compare the overall survival of patients treated with these regimens.
* Determine the safety of erlotinib in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease stage (I-II vs III-IV), participating center, age (≤ 65 vs > 65), response to first-line therapy (no evidence of disease/complete response vs partial response vs stable disease), and first-line therapy (platinum-based vs platinum/taxane combination vs platinum-based triplet). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral erlotinib once daily for up to 2 years in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo observation as per standard of care. Quality of life is assessed at baseline and then every 3 months for up to 2 years.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 830 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, primary peritoneal, or fallopian tube cancer meeting 1 of the following criteria:

  * High-risk stage I disease, as defined by grade 3, aneuploid grade 1 or 2, or clear cell disease
  * Stage II, III, or IV disease
* Completed first-line therapy within the past 6 weeks

  * Received a platinum derivative (carboplatin or cisplatin) alone or in combination with other agents for 6-9 courses
  * Must have achieved complete response/no evidence of disease, partial response, or stabilization of disease after therapy
* No adenocarcinoma of unknown origin
* No known brain metastases or leptomeningeal disease

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Platelet count ≥ 100,000/mm^3
* WBC ≥ 2,000/mm^3

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (≤ 5 times ULN in patients with known liver metastases)
* Bilirubin ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 5 times ULN except in patients with known bone metastases
* PT and PTT ≤ 1.5 times ULN

Renal

* Creatinine ≤ 2 times ULN

Cardiovascular

* No myocardial infarction within past 6 months
* No second- or third-degree heart block without pacemaker

Gastrointestinal

* No active peptic ulcer disease
* No gastrointestinal tract disease that would interfere with ability to take oral medications, affect absorption, or require parenteral nutrition
* No uncontrolled inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant dermatologic disease
* No inflammatory changes to the surface of the eye
* No history of allergic reaction to compounds of similar chemical composition as erlotinib
* No other significant medical condition or neurologic or psychiatric disorder
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or cone-biopsied carcinoma in situ of the cervix
* No psychiatric illness or familial, geographic, or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior therapy targeting epidermal growth factor receptor
* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* See Surgery
* No concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy

Radiotherapy

* No prior radiotherapy unless completed more than 5 years ago AND outside the abdomen/pelvis

Surgery

* Interval debulking surgery after 3 courses of chemotherapy and second-look surgery at the end of chemotherapy allowed as per study EORTC-55971/NCIC OV13/Chorus

Other

* No other prior or concurrent investigational agents
* No other concurrent anticancer treatment
* Concurrent participation in study EORTC-55971/NCIC-OV13/Chorus allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 835 (Actual)
Dates: Start 2005-09; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Overall survival
Adverse event profile
Quality of life
Cutaneous toxicity (rash or acne [papulo-pustular rash])

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Jimeno, Study Chair — Hospital Universitario 12 de Octubre
Locations (92):
- Australia (9):
  - Prince of Wales Private Hospital, Randwick, New South Wales
  - Tamworth Base Hospital, Tamworth, New South Wales
  - Manning Base Hospital, Taree, New South Wales
  - Newcastle Mater Misericordiae Hospital, Waratah, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Royal Women's Hospital, Carlton, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Murray Valley Private Hospital and Cancer Treatment Centre, Wodonga, Victoria
  - Sir Charles Gairdner Hospital - Nedlands, Nedlands, Western Australia
- Austria (2):
  - Landeskrankenhaus Klagenfurt, Klagenfurt
  - A.o. Bezirkskrankenhaus Kufstein, Kufstein
- France (36):
  - Centre Hospitalier de L' Agglomeration Montargoise, Amilly
  - Centre Hospitalier General, Amilly
  - Centre Hospital General Robert Ballanger, Aulnay-sous-Bois
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Clinique Tivoli, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Boucher
  - Centre Regional Francois Baclesse, Caen
  - Centre Hospitalier Regional de Chambery, Chambéry
  - Centre Jean Perrin, Clermont-Ferrand
  - Hopital Louis Pasteur, Colmar
  - Centre Hospitalier de Dax, Dax
  - Clinique Pasteur, Évreux
  - Centre Hospitalier de Gap, Gap
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Clinique Victor Hugo, Le Mans
  - Centre Hospitalier Bretagne Sud, Lorient
  - Centre Leon Berard, Lyon
  - Hopital Saint Joseph, Marseille
  - Centre Hospitalier General de Mont de Marsan, Mont-de-Marsan
  - Centre Hospitalier General Andre Boulloche, Montbéliard
  - Centre Hospitalier de Montlucon, Montluçon
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Hotel Dieu de Paris, Paris
  - Institut Curie Hopital, Paris
  - Polyclinique Francheville, Périgueux
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - Centre Paul Strauss, Strasbourg
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Centre Hospitalier Valence, Valence
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
- Italy (8):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Ospedale Sant Anna, Como
  - Ospedale Santa Maria Goretti, Latina
  - Ospedale Niguarda Ca'Granda, Milan
  - Ospedale San Gerardo, Monza
  - Universita di Torino, Turin
  - Azienda Sanitaria Ospedaliera Ordine Mauriziano, Turin
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Netherlands (6):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Martini Ziekenhuis, Groningen
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - Erasmus MC - Sophia Children's Hospital, Rotterdam
- Hospitais da Universidade de Coimbra (HUC), Coimbra, Portugal
- Spain (5):
  - Institut d'Oncologia Corachan, Barcelona
  - Hospital Universitario San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Instituto Valenciano De Oncologia, Valencia
- United Kingdom (25):
  - Stoke Mandeville Hospital, Aylesbury-Buckinghamshire, England
  - North Devon District Hospital, Barnstaple, England
  - Royal United Hospital, Bath, England
  - City Hospital - Birmingham, Birmingham, England
  - Cumberland Infirmary, Carlisle, England
  - Queen Elizabeth Hospital, Gateshead, England
  - Ipswich Hospital, Ipswich, England
  - University College Hospital, London, England
  - Mid Kent Oncology Centre at Maidstone Hospital, Maidstone, England
  - Queen Elizabeth The Queen Mother Hospital, Margate, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - St. Mary's Hospital, Newport, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Royal Preston Hospital, Preston, England
  - Royal Shrewsbury Hospital, Shrewsbury, England
  - Wexham Park Hospital, Slough, Berkshire, England
  - Southampton General Hospital, Southampton, England
  - Staffordshire General Hospital, Stafford, England
  - Yeovil District Hospital, Yeovil, England
  - Gartnavel General Hospital, Glasgow, Scotland
  - Bronglais District General Hospital, Aberystwyth, Wales
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - South West Wales Cancer Institute, Swansea, Wales

REFERENCES:
- [Derived] Vergote IB, Jimeno A, Joly F, Katsaros D, Coens C, Despierre E, Marth C, Hall M, Steer CB, Colombo N, Lesoin A, Casado A, Reinthaller A, Green J, Buck M, Ray-Coquard I, Ferrero A, Favier L, Reed NS, Cure H, Pujade-Lauraine E. Randomized phase III study of erlotinib versus observation in patients with no evidence of disease progression after first-line platin-based chemotherapy for ovarian carcinoma: a European Organisation for Research and Treatment of Cancer-Gynaecological Cancer Group, and Gynecologic Cancer Intergroup study. J Clin Oncol. 2014 Feb 1;32(4):320-6. doi: 10.1200/JCO.2013.50.5669. Epub 2013 Dec 23. PMID 24366937